CLINICAL TRIAL: NCT00750152
Title: A Phase 3 Double-Blind, Randomized, Placebo-Controlled,Multicenter, Parallel Group Evaluation of the Efficacy and Safety of NAFT-500 in Subjects With Tinea Cruris
Brief Title: Multicenter Study of the Safety and Efficacy of NAFT-500 in Tinea Cruris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRZ 90200/FI/3001
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Results first posted 2012-03-13 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2012-10

CONDITIONS: Tinea Cruris; Jock Itch
Keywords: tinea cruris; jock itch
MeSH Terms: conditions — Tinea Cruris

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator): placebo
  Interventions: Drug: Placebo
- 1 (Experimental): NAFT-500
  Interventions: Drug: NAFT-500

INTERVENTIONS:
Drug: NAFT-500 — topical cream application up to 4 weeks
  Arms: 1
Drug: Placebo — placebo cream applied for up to 4 weeks
  Arms: 2

SUMMARY:
A research study to compare the safety and effectiveness of an investigational medication called NAFT-500 to placebo (no active treatment), when used in subjects with tinea cruris, also known as jock itch.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of NAFT-500, applied once daily for 2 weeks, compared to placebo in the treatment of subjects with potassium hydroxide (KOH) and culture positive symptomatic tinea cruris.

ELIGIBILITY:
Inclusion Criteria:

1. Review and sign a statement of Informed Consent and HIPAA authorization.
2. Males or non-pregnant females ≥12 years of age, of any race or sex. Females of childbearing potential must have a negative urine pregnancy test.
3. For minors (less than 18 years), the parent/legal guardian must complete the informed consent process AND the subject must complete the assent process and sign the appropriate form (if age appropriate).
4. Presence of tinea cruris characterized by clinical evidence of a tinea infection (at least moderate erythema, moderate scaling, and mild pruritus) as confirmed by signs and symptoms.
5. KOH positive and culture positive baseline skin scrapings obtained from the site most severely affected or a representative site of the overall severity.
6. Subjects must be in good health and free from any clinically significant disease that might interfere with the study evaluations.
7. Subjects must be able to understand the requirements of the study and willing to comply with the study requirements.

Exclusion Criteria:

1. A life-threatening condition (ex. autoimmune deficiency syndrome, cancer, unstable angina, or myocardial infarction) within the last 6 months.
2. Subjects with abnormal findings - physical or laboratory - that are considered by the investigator to be clinically important and indicative of conditions that might complicate interpretation of study results.
3. Subjects with a known hypersensitivity to study medications or their components.
4. Subjects who have a recent history or who are currently known to abuse alcohol or drugs.
5. Uncontrolled diabetes mellitus.
6. Hemodialysis or chronic ambulatory peritoneal dialysis therapy.
7. Current diagnosis of immunocompromising conditions.
8. Atopic or contact dermatitis.
9. Severe dermatophytoses, mucocutaneous candidiasis, or bacterial skin infection.
10. Female subject who is pregnant or lactating, who is not using or does not agree to use an acceptable form of contraception during the study, or who intends to become pregnant during the study (females who are surgically sterilized or post menopausal for at least 2 years are not considered to be of childbearing potential). For the purposes of this study,acceptable forms of birth control include: oral contraceptives, contraceptive patches/implants, double barrier methods (e.g., use of condom and spermicide), IUD, and abstinence with second acceptable method should subject become sexually active.
11. Subjects using the following medications:

    * Topical anti-fungal therapy, powders or topical corticosteroids applied within 14 days prior to randomization. Terbinafine, butenafine, and naftifine (topical) within 30 days prior to randomization.
    * Oral anti-fungal therapies within 3 months of randomization (8 months for oral terbinafine).
    * Systemic antibiotic or corticosteroid treatment within 30 days of randomization.
    * Any other significant treatments, except hormonal contraception and multivitamin, at the discretion of the investigator that would interfere with study treatment.
    * Investigational drug/ device within 30 days of randomization

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2008-09; Primary Completion 2009-08 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Parish, MD, Principal Investigator — Paddington Testing Company
Locations (20):
- United States (15):
  - Radiant Research, Birmingham, Alabama
  - University Clinical Trials, San Diego, California
  - University of California San Francisco Dept of Dermatology, San Francisco, California
  - FXM Research, Miami, Florida
  - FXM Research, Miramar, Florida
  - Tulane Univeristy Health Services Ctr., New Orleans, Louisiana
  - Silverton Skin Institute, Grand Blanc, Michigan
  - Zoe Draelos, MD, High Point, North Carolina
  - Haber Dermatology, Euclid, Ohio
  - Paddington Testing Company, Philadelphia, Pennsylvania
  - Tennesse Clinical Research, Nashville, Tennessee
  - J&S Studies, College Station, Texas
  - Research Across America, Dallas, Texas
  - Research Across America, Plano, Texas
  - Oakwell Clinical Research, San Antonio, Texas
- Puerto Rico (5):
  - Edwin Camilio Vazquez, MD, Aguas Buenas
  - Medicina General y Cirugia Menor, Cayey
  - Advanced Medical Concepts, PSC, Cidra
  - Manuel Guzman, MD, Humacao
  - Isabel Quijano, MD, Rio Piedras

REFERENCES:
- [Result] Parish LC, Parish JL, Routh HB, Avakian E, Olayinka B, Pappert EJ, Plaum S, Fleischer AB, Hardas B. A double-blind, randomized, vehicle-controlled study evaluating the efficacy and safety of naftifine 2% cream in tinea cruris. J Drugs Dermatol. 2011 Oct;10(10):1142-7. PMID 21968664
- See also: Naftin Cream 2% product information — http://dailymed.nlm.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- NAFT-500: Naftin 2% cream applied daily for 2 weeks
- Placebo-2wks: Placebo cream applied daily for 2 weeks
Period: Overall Study
Arm/Group | NAFT-500 | Placebo-2wks
Started | 166 | 168
Completed | 144 | 141
Not Completed | 22 | 27
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 8 | 13
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Physician Decision | 1 | 1
Not completed — Non-compliance | 0 | 1
Not completed — Termination by sponsor | 1 | 0
Not completed — Other | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NAFT-500 | Placebo-2wks | Total
Number analyzed (Participants) | 166 | 168 | 334
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 0 | 4
  Between 18 and 65 years | 139 | 149 | 288
  >=65 years | 23 | 19 | 42
Age Continuous [Mean (Standard Deviation); unit: years] | 47.2 (15.54) | 46.2 (14.53) | 46.7 (15.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 30 | 52
  Male | 144 | 138 | 282
Region of Enrollment [Number; unit: participants]
  United States | 112 | 113 | 225
  Puerto Rico | 54 | 55 | 109

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects
Description: Complete cure is defined as negative mycology results from the central laboratory (dermatophyte culture and KOH) and absence of Erythema, Scaling, and Pruritus (grade 0 for each) evaluated using the 5-point severity grading scale: 0 = absent, 1 = mild, 2 = moderate, 3 = marked, and 4 = not done.
Time Frame: Week 4 post-baseline
Population: The Full Analysis Set (FAS)is the subset of all subjects in the Safety Evaluation Set (SES)with a positive culture at baseline and for whom the primary efficacy variable is available. This is a modified intent-to-treat (MITT) principle because the culture results were not available before the start of treatment.
Measure: Number; unit: percentage of subjects with complete cur
Arm/Group | NAFT-500 | Placebo-2wks
Number analyzed (Participants) | 75 | 71
percentage of subjects with complete cur | 25.3 | 2.8
Statistical Analysis 1: Comparison: NAFT-500 vs Placebo-2wks; In order to compare complete cure rate in the NAFT-500 group with that in the placebo group, the following one-sided null and alternate hypotheses will be tested: * H0: p1 <= p0 * Ha: p1 > p0 where p0 and p1 denote the proportion of subjects with complete cure in the placebo and NAFT-500 groups, respectively; Test type: Superiority or Other; p = 0.025, Cochran-Mantel-Haenszel; The CMH test after stratification by site compared the proportion of complete cure in NAFT-500 to that of placebo to evaluate its superiority; one-sided p-value from CMH test = 0.001

2. Secondary Outcome: Mycological Cure and Treatment Effectiveness
Description: Mycological Cure was defined as negative KOH result and negative dermatophyte culture at Week 4. Treatment Effectiveness as defined as negative KOH, negative culture, and Scaling, Erythema and Pruritis grades of 0 or 1 at Week 4.
Time Frame: Week 4 (two weeks post-treatment)
Population: This is the Full Analysis Set (FAS)comprising of subjects in the SES with a positive culture at Baseline for whom the primary efficacy variable was available. This was a modified intent to treat principle because the culture results were not available before the start of treatment.
Measure: Number; unit: percentage of subjects
Arm/Group | NAFT-500 | Placebo-2wks
Number analyzed (Participants) | 75 | 71
percentage of subjects
  Mycological Cure (MC) | 72.0 | 15.5
  Treatment Effectiveness (TE) | 60.0 | 9.9

ADVERSE EVENTS:
Arm/Group | NAFT-500 | Placebo-2wks
Serious Adverse Events (participants affected / at risk) | 0/166 | 0/168
Other Adverse Events (participants affected / at risk) | 4/166 | 10/168
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NAFT-500 (N=166) | Placebo-2wks (N=168)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 4
Headache (Nervous system disorders) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Principal Investigator agree not to individually publish the results of the Study. Institution and Principal Investigator may, however, upon written notice to Merz participate in a joint, multicenter publication of the Study results with other investigators and/or institutions, provided that the manuscript or abstract is first reviewed by Merz.